CLINICAL TRIAL: NCT00951366
Title: Preterm Lung Patient Registry
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Lystra Hayden, Instructor in Pediatrics, Boston Children's Hospital
Other Study IDs: X08-07-0335
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Bronchopulmonary Disease
Keywords: premature birth; neonatal respiratory distress; chronic lung disease; epidemiologicfactors; genetic factors
MeSH Terms: conditions — Premature Birth; Pulmonary Atelectasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 21 Years
Biospecimen Retention: Samples With DNA — Buccal swabs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bronchopulmonary Dysplasia (BPD)
  Interventions: Other: Patient Registry

INTERVENTIONS:
Other: Patient Registry — The CHILD Clinic Patient Registry is an observational study designed to identify epidemiologic and genetic factors associated with chronic lung disease in former preterm infants or those with lung disease in the neonatal period.

SUMMARY:
The goal of the Preterm Lung Patient Registry is to collect data on individuals with neonatal lung disease to better understand the illness and ultimately improve their care and survival. The Patient Registry was established in 2008 as a means to monitor important trends in the BPD population and to improve understanding, treatment, and survival.

DETAILED DESCRIPTION:
The Preterm Lung Patient Registry is an observational study designed to identify epidemiologic and genetic factors associated with chronic lung disease in former preterm infants or those with lung disease in the neonatal period. The Patient Registry is used by both clinicians and researchers to better understand BPD and to improve care of individuals with BPD. It is used to assess phenotype and genotype information from former preterm infants with lung disease. Data in the Patient Registry will be analyzed and an regular report of BPD health trends will be created. Using this information, BPD clinicians can address quality improvement initiatives, and examine changing health care issues, including nutritional status, infection control, pulmonary treatment, metabolic and associated genetic variants. The Patient Registry will also play an important role in directing clinical care and in the design of clinical research studies. Researchers use the registry to help in investigating various aspects of neonatal lung diseases like BPD, including medications, diagnostic procedures, and eligibility for clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Former preterm infant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Former preterm infants
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2008-06 (Actual); Primary Completion 2099-01-01 (Estimated); Study Completion 2099-01-01 (Estimated)

PRIMARY OUTCOMES:
Lung function | Lifetime
  Spirometry

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Annesi CA, Levin JC, Litt JS, Sheils CA, Hayden LP. Long-term respiratory and developmental outcomes in children with bronchopulmonary dysplasia and history of tracheostomy. J Perinatol. 2021 Nov;41(11):2645-2650. doi: 10.1038/s41372-021-01144-0. Epub 2021 Jul 21. PMID 34290373
- [Result] Levin JC, Sheils CA, Gaffin JM, Hersh CP, Rhein LM, Hayden LP. Lung function trajectories in children with post-prematurity respiratory disease: identifying risk factors for abnormal growth. Respir Res. 2021 May 10;22(1):143. doi: 10.1186/s12931-021-01720-0. PMID 33971884